CLINICAL TRIAL: NCT02124941
Title: Glutamate-Glutamine Cycling (VCYC) During Cocaine Abstinence Using 1H-MRS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1311013082; 1R21DA044005-01 (NIH); 1R21DA043055-01 (NIH)
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Cocaine Dependence; Healthy
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

ARMS (4):
- 1H MRS (Experimental): All subjects will undergo three magnetic resonance spectroscopy (1H-MRS) scans, including before and after two-weeks of placebo and NAC administration.
  Interventions: Diagnostic Test: 1H MRS
- [18F]-FDG PET scan (Experimental): All subjects will undergo [18F]FDG PET to establish previously demonstrated reductions in glucose utilization in PFC and assess VS/nucleus accumbent metabolism at baseline.
  Interventions: Diagnostic Test: [18F]FDG PET scan
- [11C]APP311 PET scan (Experimental): All subjects will undergo [11C]APP311 PET imaging to investigate whether there are differences in synaptic integrity / neuronal plasticity in the brains of individuals abstinent from cocaine compared to healthy controls at baseline.
  Interventions: Diagnostic Test: [11C]APP311 PET scan
- Medication (NAC & placebo) administration (Active Comparator): Upon completion of baseline (abstinence) 1H-MRS scanning at 7T, CU and HC subjects will participate in two additional 1H-MRS scans, including after 2 weeks of placebo and 2 weeks of NAC administration (3600 mg/day) given in double-blind, randomized, counterbalanced order.
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — Upon completion of baseline (abstinence) 1H-MRS scanning, CU and HC subjects will participate in two additional 1H-MRS scans, including after 2 weeks of placebo and 2 weeks of NAC administration (3600 mg/day) given in double-blind, randomized, counterbalanced order.
  Arms: Medication (NAC & placebo) administration
Diagnostic Test: [18F]FDG PET scan — All subjects will undergo [18F]FDG PET to establish previously demonstrated reductions in glucose utilization in PFC and assess VS/nucleus accumbent metabolism at baseline.
  Arms: [18F]-FDG PET scan
Diagnostic Test: 1H MRS — All subjects will undergo three magnetic resonance spectroscopy (1H-MRS) scans at 7T, including before and after two-weeks of placebo and NAC administration.
  Arms: 1H MRS
Diagnostic Test: [11C]APP311 PET scan — All subjects will undergo [11C]APP311 PET imaging to investigate whether there are differences in synaptic integrity / neuronal plasticity in the brains of individuals abstinent from cocaine compared to healthy controls at baseline.
  Arms: [11C]APP311 PET scan

SUMMARY:
This study is designed to look at the relationship between brain glucose utilization, neurotransmission (e.g., glutamate, also known as the main excitatory amino-acid neurotransmitter in the brain), and synaptic density. This relationship will be explored in the brain's prefrontal cortex, an area important in decision-making and impulsivity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years;
2. Voluntary, written, informed consent;
3. Physically healthy by medical history, physical, neurological, ECG and laboratory examinations;
4. DSM-IV criteria for Cocaine Dependence (304.20) (Note: subjects will also meet DSM-5 criteria for Cocaine Use Disorder);
5. Documented evidence (by urine toxicology) of abstinence from cocaine (2 weeks for scan 1, and 2 and 4 weeks for scans 2 and 3, respectively)
6. Full scale and verbal IQs > 80;
7. For females, a negative serum pregnancy test (β-HCG) at screening and negative urine pregnancy test on PET scan day prior to imaging.

Exclusion Criteria:

1. A history of other substance dependence (e.g., alcohol, opiates, sedative hypnotics), except for nicotine;
2. A primary DSM-IV Axis I major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the Structured Clinical Interview for DSM-IV (SCID);
3. A history of significant medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular, seizure, traumatic brain injury) illness;
4. Current use of psychotropic and/or potentially psychoactive prescription medications;
5. Medical contraindications to participation in a magnetic resonance imaging procedure (e.g., ferromagnetic implants/foreign bodies, claustrophobia, cardiac pacemaker, prosthetic valve, otologic implant, etc.);
6. For females, laboratory (β-HCG) evidence of pregnancy, physical evidence of pregnancy;
7. For subjects interested in pharmacotherapy component, history of allergies to NAC and current elevation on liver function tests above twice the normal limit;
8. Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year;
9. Subjects with current, past or anticipated exposure to radiation in the work place within one year of proposed research PET scans;
10. History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto);
11. Blood donation within eight weeks of the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
GLU and GLU/GLN ratios | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Angarita, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States